CLINICAL TRIAL: NCT05296889
Title: Multicenter Post-Market Clinical Follow-Up Study on the Safety and Performance of Ennovate® Cervical - a Prospective Study on Total Indications
Brief Title: Post-Market Clinical Follow-Up Study on the Safety and Performance of Ennovate® Cervical
Acronym: CERISE
Status: Recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: Raylytic GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2010
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Spine Fracture; Degenerative Disc Disease; Spinal Instability; Spinal Tumor; Degenerative Myelopathy
Keywords: Cervical Spine
MeSH Terms: conditions — Spinal Fractures; Intervertebral Disc Degeneration; Spinal Cord Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ennovate® Cervical: Alll patients which were treated with the Ennovate® Cervical system in accordance with the indications given in the instructions for use
  Interventions: Device: posterior stabilization for the cervical spine

INTERVENTIONS:
Device: posterior stabilization for the cervical spine — The Ennovate® Cervical Spinal System is a posterior stabilization for the cervical and upper-thoracic spine. The implants are used for the posterior monosegmental and multisegmental stabilization of the occipitocervical junction and of the cervical and upper thoracic spine.

SUMMARY:
Multicenter Post market clinical follow-up Study on the Safety and Performance of Ennovate® Cervical - Prospective, pure data collection of all Ennovate Cervical patients in Total Indications

DETAILED DESCRIPTION:
This clinical study is one of the Post market clinical follow-up measures that enables the manufacturer to monitor the clinical safety and performance of the Ennovate® Cervical system. The study enables a quick, but detailed implant documentation, which is of great interest for the current and future users of the internal fixation system targeted in this study. It includes the relevant outcomes to evaluate safety and efficacy of the implant system for various indications in trauma and degenerative disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patient is minimum 18 years old
* Informed Consent in the documentation of clinical and radiological results
* Patient has indication according to Instructions for Use (IFU)
* Patient is not pregnant

Exclusion Criteria:

* Patient's clear unability or unwillingness to participate in follow-up examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated with the Ennovate® Cervical system in accordance with the indications given in the instructions for use: fractures, degenerative instability, post-trauma instability, tumors, degenerative cervical myelopathy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change of Pain | preoperatively, at 3 months postoperatively and at 12 months postoperatively
  Pain will be assessed by the patient using the Visual Analogue Scale (VAS) which states "0" at one end representing "no pain" and "100" at the opposite end representing "maximal/worst pain".

SECONDARY OUTCOMES:
Change of Quality of life | preoperatively, at 3 months postoperatively and at 12 months postoperatively
  In order to analyze the quality of life of the patients, the 5-dimension 5-level score of EuroQol Group (EQ-5D-5L) is used. The score is self-completed by the patient. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Change of Neurological status | preoperatively, at 3 months postoperatively and at 12 months postoperatively
  The Japanese Orthopaedic Association (JOA) myelopathy score is a disease-specific and physician oriented system that mainly assesses the neurological status of the patient and enables surgeons to compare the changes in the neurological status of the patient before and after certain treatments. However, the JOA score does not include patients' satisfaction, disability, handicaps, or general health (physical and mental health), which can be affected by cervical myelopathy.
Change of Disability | preoperatively, at 3 months postoperatively and at 12 months postoperatively
  The Neck Disability Index (NDI) is designed to measure neck-specific disability. The questionnaire has 10 items to measure patient-reported disability secondary to neck pain and activities of daily living including personal care, lifting, reading, headaches, concentration, work status, driving, sleeping and recreation and patients rate their status from 0 (best) to 5 (worst imaginable). Individual item responses are summed to a total score, where 0 points indicate no activity limitations and 50 points indicate complete activity limitation.
Bone fusion | at final follow-up 12 months postoperatively
  After cervical stabilization fusion of the treated segment is aspired in most cases. The fusion status can be determined from radiographs (static or dynamic). Bony fusion can be characterized quantitatively by the fusion rate.
Cumulative number of side effects | throughout the follow-up up to 12 months postoperatively
  Occurrence of complications potentially associated with the implanted devices can never be fully excluded during spinal surgery. In order to monitor potential complication and to identify so far unknown complications Adverse Events and Serious Adverse Events deemed related to the investigational device are recorded.

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Krankenhaus Ludmillenstift Meppen, Meppen, Lower Saxony
  - Städtisches Klinikum Dresden, Dresden, Saxony
  - Berufsgenossenschaft Klinikum Bergmannstrost Halle / Saale, Halle, Saxony-Anhalt
  - Schön Klinik Hamburg Eilbek, Hamburg

IPD SHARING:
Plan to Share IPD: No